CLINICAL TRIAL: NCT03387254
Title: Virtual Reality and Brain Stimulation, an Experiential Approach
Acronym: REVISTIM-X
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: RC17_0174
Record Dates: First submitted 2017-11-24; First posted 2018-01-02 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Acrophobia
Keywords: virtual reality; brain stimulation
MeSH Terms: conditions — Acrophobia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR + active brain stimulation (Experimental): Exposure to a virtual reality world with active transcranial electric stimulation
  Interventions: Device: VR + active brain stimulation
- VR + sham brain stimulation (Sham Comparator): Exposure to a virtual reality world with sham transcranial electric stimulation
  Interventions: Device: VR + sham brain stimulation

INTERVENTIONS:
Device: VR + active brain stimulation — Active Brain stimulation (tDCS) is applied during exposition to virtual reality (20 minutes)
  Arms: VR + active brain stimulation
Device: VR + sham brain stimulation — Sham Brain stimulation (tDCS) is applied during exposition to virtual reality (20 minutes)
  Arms: VR + sham brain stimulation

SUMMARY:
The aim of this study is to assess feasibility, acceptability and efficacy of two VRET (Virtual Reality Exposition Therapy)session associated with either active anodal tDCS or sham tDCS on the ventromedial prefrontal cortex to decrease anxiety related to visual height intolerance

DETAILED DESCRIPTION:
Subjects suffering from visual height intolerance are asked to go in 20 min as height as possible riding in two elevators of adjacents buildings separated by a board they have to cross at each stage.

Inclusion visit:

* Confirmation of eligibility criteria
* Written informed consent
* Completion of Acrophobia Questionnaire (AQ), Attitude towards Height Questionnaire (ATHQ), Height Interpretation Questionnaire (HIQ), Visual Height Intolerance scale(vHI), State-Trait Anxiety (STAI), Inventory and Clinical Global Impressions (CGI)
* Virtual task (10 minutes): riding in an elevator. At each level,subjects are asked to rate their Subjective Units Discomfort (SUD scale from 0 to 100).
* Assessment of basal cortisol before beginning of exposure to virtual reality (sampling saliva through a Salivette®)
* Pulse and blood pressure measurements before and after session

Session 1 (within 1 to 7 days following Inclusion Visit) and session 2 (within 48 hours following session 1):

* Randomization is made by the tDCS software (double bind).
* Equipment of subject with Vive Headset (virtual reality HTC vive), trackers and (tDCS). The subject does not see the experimental room.
* Virtual task (20 minutes): the subject has to ride in an elevator up to the next floor, cross a footbridge between 2 buildings to access the elevator on the other side and be able to climb to the next floor. At each level, the subject asked to rate their SUD. The objective is to climb as high as possible.
* The active or sham brain stimulation is applied randomly during the entire virtual task.
* Assessment of basal cortisol before and after exposure to virtual reality
* Pulse and blood pressure measurements before and after session
* After session: debriefing and explication of the subjective experience (30 minutes).

End of study visit:

* Identical to inclusion visit plus :
* acrophobia/visual height
* Completion of Simulator Sickness Questionnaire (SSQ) and Igroup Presence Questionnaire (IPQ)

ELIGIBILITY:
Inclusion Criteria:

* Without any particular ethnic and psychosocial criteria
* Subjects with fear of heights (anxiety AQ score >45 and/or VHI score >7)
* Subjects with SUD score>50/100 assessed during first visit
* Subjects without psychiatric or addictive disorders
* Subjects without criteria of phobia according to DSM5 (Diagnostic Statistical Manual)

Exclusion Criteria:

* contraindication to tDCS (neurosurgical history, intracranial device, skin problems)
* current virtual reality intolerance
* history of psychiatric or addictive disorders
* Use of psychotropic drugs
* Use of non psychotropic treatments significantly influencing mood or level of anxiety
* Neurological pathology, locomotor disability, or sensory (vestibular, visual, auditory ...)
* pregnant or breast-feeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2018-07-27 (Actual)

PRIMARY OUTCOMES:
Change in Subjective Units of Discomfort (SUD) at different heights | within 2 weeks
  Measure by 0 to 100 scale (100 being the most intense fear) subjective units of discomfort of subjects at different heights (corresponding to virtual floor of a flat) and at each visit

SECONDARY OUTCOMES:
Change in composite score of Stress reactivity and intolerance of heights | within one week
  Evaluated by psychometric questionnaires : Acrophobia Questionnaire (AQ), Attitude towards Height Questionnaire (ATHQ), Height Interpretation Questionnaire (HIQ), Visual Height Intolerance scale(vHI), State-Trait Anxiety (STAI), Inventory and Clinical Global Impressions (CGI)
  The results of these questionnaires will be computed to obtain an overall assessment of the change in reactivity to stress.
  Comparison of results between the 2 arms
Change in physiologic effects | within 2 weeks
  Evaluation of physiologic effects by skin conductance, pulse, salivary cortisol level, eye-tracking.
  The results of these exams and measures will be computed to obtain an overall assessment of the change in physiologic effects at each visit
Comparison in composite score of performance in virtual reality | within 2 weeks
  Assessing the performances in virtual reality in both groups at inclusion and endpoints visits, evaluated by
  * height and number of floor achieved
  * rating of SUD at each floor
  * time spent at each floor
  * Differences in eye behavior (duration of fixations, saccade length ...) and in the deployment of visual attention
Debriefing | within one week
  Analysis after sessions of subjective experience and acceptability using explicationy interviews based on micro phenomenology Locating some recurrences and particularity in the phenomenological experience of patients according to the different experimental conditions.
Quality of immersion | at 2 weeks
  Measured by the score to the Igroup Presence Questionnaire
virtual reality and tDCS tolerance | at 2 weeks
  Measured by the Simulator sickness questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Nantes, France